CLINICAL TRIAL: NCT05557539
Title: Hypothesizing the Genesis of Infectious Diseases and Epidemics Through an Integrated Systems Biology Approach
Acronym: HYGIEIA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2021/30DEC/543
Record Dates: First submitted 2022-09-23; First posted 2022-09-28 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: SARS-CoV-2 Infection; Influenza Viral Infections
MeSH Terms: conditions — COVID-19 | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- all patients (Other): The intervention consists of taking blood samples, urine sample and naso-pharyngeal sample at two different time points (at inclusion and at week8-12).
  Interventions: Biological: blood samples, urine samples and nasopharyngeal swabs

INTERVENTIONS:
Biological: blood samples, urine samples and nasopharyngeal swabs — The following samples will be collected: First time point : 6 blood sample tubes (5mL EDTA, 5mL heparinized and 7.5mL heparinized, 5mL citrate, 5mL serum, 5mL Tempus Blood RNA Tube); 1 urine sample (10mL in a sterile collector) and 1 naso-pharyngeal swab (1mL UT medium). Second time point : 5 blood sample tubes (5mL EDTA,5mL heparinized and 7.5mL heparinized, 5mL serum, 5mL Tempus Blood RNA Tube); 1 urine sample (10mL in a sterile collector) and 1 naso-pharyngeal swab (1mL UT medium).

SUMMARY:
In this study, the investigators aim to collect phenotypical and extensive unbiased multimodal biological data, at two different time points, and to integrate them using a systems biology approach.

The present project aims at generating a systems biology network that can recapitulate the complexity of processes underlying differential SARS-CoV-2 phenotypic responses through exploitation of clinical -omics data. Identifying key determinants and mechanisms of biological variability responsible for phenotypic differences will lead to a better management of patients through the application of precision medicine.

DETAILED DESCRIPTION:
HYGIEIA is a multicentric prospective interventional study. The study has two parts, Part 1 with prospective data and sampling, and Part 2 based on samples that were previously collected and stored within COBISA study (2020/11MAI/269).

i. In Part 1, patients acutely infected with SARS-COV-2 will be proposed inclusion. Included patients will be sampled at two different time points (acute infection and convalescent phase, i.e. 8-12 weeks later). Samples will be analysed using cutting edge -omics technologies in order to characterize the genotypic, proteomic, transcriptomic, metabolomic and respiratory microbiota/virome profile through explorative approaches. Clinical and routine biological data will be prospectively collected either as outpatients or during the acute hospitalization and convalescent phase.

ii. In Part 2, samples collected and biobanked during the COBISA study (2020/11MAI/269) will be analysed similarly to the samples collected during the prospective part. Clinical and routine biological data will be retrospectively collected using the patients electronic medical record (EMR).

Generated data will be integrated using a systems biology approach with algorithms developed by a biostatistics team.

ELIGIBILITY:
Inclusion Criteria:

* For all: (1) 18 years or over; (2) Patient or legal representative have provided informed consent.
* Cases: Reverse-transcriptase polymerase chain reaction (RT-PCR) confirmed symptomatic SARS-CoV-2 infection.
* Controls :

  1. Patient presenting with acute respiratory failure: (1) Patient presenting with hypoxemic respiratory failure diagnosed by the treating physician and influenza proven as the cause of the respiratory failure; (2) active SARS-CoV-2 infection excluded by RT-PCR and deemed non-probable by the treating physician.
  2. Healthy controls : (1) Patients presenting without acute respiratory failure (ie. SpO2 >93%); (2) no RT-PCR or antigen rapid test proven SARS-CoV-2 infection within the last 6 months; (3) no active respiratory tract infection.
  3. Dexamethasone controls: Patient presenting to the day hospital for an upper or lower limb surgery and who will receive dexamethasone in this context. The criteria for healthy controls also apply.

Exclusion Criteria:

* For all: (1) <18 years old ; (2)unwilling to provide informed consent; (3) pregnancy at the time of inclusion
* For cases: Asymptomatic infection
* For controls:

  1. Active COVID-19 infection diagnosed by RT-PCR or suspect according to the treating physician at the time of inclusion,
  2. For healthy controls: Acute or chronic respiratory failure.
  3. Patient currently receiving dexamethasone (i.e. before study inclusion). The criteria for healthy controls also apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 249 (Actual)
Dates: Start 2022-02-07 (Actual); Primary Completion 2024-12-18 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Change on the 11 points World Health Organization (WHO) clinical progression scale | At inclusion (for hospitalized patients daily evaluation untill discharge) and at the end of study visit between 8 and 12 weeks later
  Evaluation of disease state on the 11 points WHO Clinical Progression Scale. The minimum value is 0 and corresponds to an uninfected status and the maximum value is 10 in case of death. So a higher score means a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Jean Cyr Yombi, MD, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (1):
- Cliniques Universitaires Saint-Luc, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No